CLINICAL TRIAL: NCT06217276
Title: Examining the Relationship Between Respiratory Muscle Fatigue and Lower Extremity Muscle Oxygenation in Chronic Obstructive Pulmonary Disease Patients.
Brief Title: Respiratory Muscle Fatigue and Lower Extremity Muscle Oxygenation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Respiratory muscle fatigue&VL
Record Dates: First submitted 2023-12-30; First posted 2024-01-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD Group (Active Comparator)
  Interventions: Other: Respiratory muscle fatigue protocol
- Healthy Group (Active Comparator)
  Interventions: Other: Respiratory muscle fatigue protocol

INTERVENTIONS:
Other: Respiratory muscle fatigue protocol — It will be performed using a powerbreath device at 60% of the maximum inspiratory pressure (MIP) amount obtained by measuring mouth pressure. The protocol includes 7 sets consisting of 2 minutes of inspiratory effort and 1 minute of rest. To further confirm the occurrence of fatigue, the patient will score fatigue using the modified Borg scale, and the score will be 5 or above11. During the application, heart rate, blood pressure and peripheral oxygen saturation will be monitored. The measurement will be performed once for each case.

SUMMARY:
In our study, changes in vastus lateralis muscle oxygenation will be evaluated with the Moxy device, a functional infrared oxygen measurement device, during the inspiratory muscle fatigue protocol in COPD cases and the healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Stage 2-3 COPD according to the following clinical diagnostic criteria according to the American Thoracic and European Respiratory Societies (ATS-ERS).
* Having been using the same medications for the last 4 weeks

Exclusion Criteria:

* Patients with severe comorbid diseases, unstable coronary artery disease, collagen vascular diseases and requiring high-flow oxygen therapy (˃ 3-4 L\min).
* Presence of any vascular problem that may affect lower extremity muscle oxygenation
* Presence of another respiratory system disease other than COPD
* Patients who have had an acute COPD exacerbation in the last 4 weeks
* Patients experiencing COPD exacerbations during the study protocol
* Presence of fatty tissue or scar tissue at the measurement points, which may impair the measurement quality.
* Have already participated in another clinical trial within the last 30 days that may affect the results of the study.

Inclusion Criteria for Healthy Cases

* Being over 18 years of age
* Not having any diagnosed chronic disease
* Not being a smoker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Lower extremity muscle oxygenation level measurement | 20 minutes
  Near Infrared Reflection Spectroscopy device will be used. The device measures and monitors muscle oxygen by taking the reflected rays of infrared rays given to the body from two different sensors to measure muscle oxygenation levels in muscle tissue. The measurement will be made in the dominant lower extremity, and the device will be placed in the mid-thigh region at the distance between the spina iliaca anterior superior reference point and the midpoint of the patella.
Lower extremity muscle total hemoglobin amount level measurement | 20 minutes
  Near Infrared Reflection Spectroscopy device will be used. The device measures and monitors muscle total hemoglobin amount by taking the reflected rays of infrared rays given to the body from two different sensors to measure muscle oxygenation levels in muscle tissue. The measurement will be made in the dominant lower extremity, and the device will be placed in the mid-thigh region at the distance between the spina iliaca anterior superior reference point and the midpoint of the patella.

SECONDARY OUTCOMES:
Peripheral oxygen saturation measurement | 20 minutes
  During the fatigue protocol, it will be measured with a finger pulse oximeter attached to the finger
Forced vital capacity (FVC), | 5 minutes
  Pulmonary function test will perform by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines. FVC is the volume of air that can forcibly be blown out after full inspiration.
Respiratory muscle strength | 10 minutes
  The mouth pressure measurement (maximum inspiratory and expiratory pressure) will perform with the Pony Fx spirometry device. Patient will place a rubber mouthpiece with flanges, on the device, exhale/inhale slowly and completely, and then will try to breath in as hard as possible. The patient will allow to rest for about a minute and the maneuver will repeat. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value will obtain.
Forced expiratory volum in one second (FEV1) | 5 minutes
  Pulmonary function test will perform by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines. FEV1 is the volume of air that can forcibly be blown out in first 1-second, after full inspiration

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided